CLINICAL TRIAL: NCT06985459
Title: Effectiveness of Exercise Relative Motion Orthoses for Improving Limited Proximal Phalangeal Joint Motion: A Single-Center, Single-Blinded Randomized Controlled Trial
Brief Title: Effectiveness of Exercise Relative Motion Orthoses for Limited Finger Joint Motion
Acronym: Exercise RM-O
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Bernadette Tobler, Head of hand therapy research unit, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM Orthosis Study 2025-00427
Record Dates: First submitted 2025-04-30; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Proximal Interphalangeal Joint Stiffness
Keywords: Proximal Interphalangeal Joint; Limited Range of Motion; Exercise Relative Motion Orthosis; Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: The investigators plan to stratify participants into two groups based on their greater PIPJ movement deficit (in flexion or in extension). Within each group, they are randomized to one of the orthosis interventions.
  This trial has four intervention arms:
  * Arm 1: PIP extension deficit treated with an exercise RMF orthosis.
  * Arm 2: PIP extension deficit treated with a placebo RMF orthosis.
  * Arm 3: PIP flexion deficits treated with an exercise RME orthosis.
  * Arm 4: PIP flexion deficits treated with a placebo RMF orthosis.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PIP extension deficit treated with an exercise RMF orthosis (Experimental): The orthosis is worn for 4 weeks. At week 6 and 8, follow-up visits are planned to measure PIPJ range of motion and patient satisfaction. For all arms, standard hand therapy treatment continues as needed.
  Interventions: Device: PIP extension deficit treated with an exercise RMF orthosis
- PIP extension deficit treated with a placebo RMF orthosis (Placebo Comparator): The orthosis is worn for 4 weeks. At week 6 and 8, follow-up visits are planned to measure PIPJ range of motion and patient satisfaction. For all arms, standard hand therapy treatment continues as needed.
  Interventions: Device: PIP extension deficit treated with a placebo RMF orthosis
- PIP flexion deficits treated with an exercise RME orthosis (Active Comparator): The orthosis is worn for 4 weeks. At week 6 and 8, follow-up visits are planned to measure PIPJ range of motion and patient satisfaction. For all arms, standard hand therapy treatment continues as needed.
  Interventions: Device: PIP flexion deficits treated with an exercise RME orthosis
- PIP flexion deficits treated with a placebo RMF orthosis (Placebo Comparator): The orthosis is worn for 4 weeks. At week 6 and 8, follow-up visits are planned to measure PIPJ range of motion and patient satisfaction. For all arms, standard hand therapy treatment continues as needed
  Interventions: Device: PIP flexion deficits treated with a placebo RMF orthosis

INTERVENTIONS:
Device: PIP extension deficit treated with an exercise RMF orthosis — The RM orthoses will be worn between 6-12 hours per day during functional use.
  Arms: PIP extension deficit treated with an exercise RMF orthosis
Device: PIP extension deficit treated with a placebo RMF orthosis — The placebo orthosis has the same design as the exercise RM orthoses, but without a difference in the extension or flexion angle, respectively, to the adjacent finger - therefore neutralizing the "quadriga phenomena", which is the effect that makes RM orthoses work.
  Arms: PIP extension deficit treated with a placebo RMF orthosis
Device: PIP flexion deficits treated with a placebo RMF orthosis — The placebo orthosis have the same design as the exercise RM orthoses, but without a difference in the extension or flexion angle, respectively, to the adjacent finger - therefore neutralizing the "quadriga phenomena", which is the effect that makes RM orthoses work.
  Arms: PIP flexion deficits treated with a placebo RMF orthosis
Device: PIP flexion deficits treated with an exercise RME orthosis — The dedicated orthosis wearing time is 6-12 hours per day during functional use.
  Arms: PIP flexion deficits treated with an exercise RME orthosis

SUMMARY:
This randomized controlled trial investigates the effectiveness of two exercise orthosis designs-the Relative Motion Flexion (RMF) and Relative Motion Extension (RME) orthoses-for improving motion in patients with proximal interphalangeal joint (PIPJ) flexion or extension deficits. A total of 148 adult patients with acute hand injuries and a minimum 10° difference between active and passive PIP joint motion will be enrolled. Participants are stratified by their primary motion deficit and randomized to either the exercise orthosis or placebo orthosis group. The orthosis is worn for 4 weeks, with follow-up assessments at weeks 6 and 8 to evaluate range of motion and patient satisfaction. All participants will continue standard hand therapy throughout the study.

DETAILED DESCRIPTION:
The prevention and treatment of proximal interphalangeal joint (PIPJ) contractures are key goals in hand rehabilitation, often addressed with orthotic interventions. The choice of orthosis design depends on the severity and timing of the injury or disease. During the acute stage, static splinting is typically used, while more dynamic orthoses, such as static-progressive splinting, are recommended in the chronic stages to manage contractures. If a contracture already exists, hand therapists differentiate between dynamic and fixed deformities in PIPJ flexion or extension. Fixed deformities do not or hardly respond to passive mobilisation, while dynamic deformities show a difference in active and passive range of PIPJ motion - e.g. in cases of soft tissue adhesions hindering active motion.

In addition to traditional passive orthoses, which stretch the PIPJ in a fixed position during dedicated periods, exercise-based orthoses (relative motion orthoses, RM) have been developed to enhance PIPJ mobility during everyday activities. These include Relative Motion Extension (RME) and Relative Motion Flexion (RMF) orthoses, designed to improve both flexion and extension. Studies have shown that RME orthoses improve active flexion, while RMF orthoses aid in active extension, with patients reporting high satisfaction and functional benefits from using these devices in daily tasks. Furthermore, RM orthoses have been widely adopted by therapists, demonstrating benefits in improving functional hand use and promoting non-intentional exercise.

Since the use of relative motion (RM) orthoses - especially as exercise orthoses - is relatively new, few prospective studies have examined their effectiveness in improving PIPJ motion. Therefore, this study aims to compare the effectiveness of exercise RM orthoses with a placebo orthosis to identify the most beneficial treatment strategies for patients with limited PIPJ motion. The goal is to strengthen the evidence base and refining the clinical application of exercise-based orthotic interventions.

The primary objective of this study is to compare the effectiveness of two orthoses designs, the exercise RME and RMF orthosis vs. a placebo orthosis.

Secondary objectives are:

1. To evaluate if there is a clinically relevant difference in activity performance at 4 and 8 weeks after orthosis fabrication.
2. To assess if there is a statistically significant difference in patient satisfaction with (i) the orthosis and (ii) treatment outcome (satisfaction with the daily use of the hand) after 4 weeks (i and ii) and 8 weeks (ii).
3. To document adherence to orthotic intervention from baseline to 4 weeks. We strive for 37 patients per arm and a total sample size of 74 patients per study group. This results in 74 patients in the extension-group and 74 patients in the flexion-group and a total of 148 patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* PIPJ motion deficit with a minimum difference of 10° between passive and active motion
* To have an acute injury, i.e. operated on or within maximum 6 weeks of accident
* Only one hand is affected
* Adult patients over 18 years of age
* Understanding German, French or English
* Hand therapy treatment in-house at Inselspital in Bern
* Ability to give informed consent as documented by signature

Exclusion Criteria:

* Previous injuries to the hand or PIPJ (e.g., intra-articular fractures, PIPJ ligament damage) that may limit baseline joint mobility and influence responsiveness to the intervention.
* Presence of conditions such as osteoarthritis (OA) or rheumatoid arthritis (RA) that may affect PIPJ stiffness, pain, or inflammation.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* Boutonniere deformity
* Minors (below 18 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Finger range of motion | Change from baseline to 2, 4 and 6 weeks
  PIPJ active and passive motion will be measured using a hand-held goniometer. The goniometer is placed dorsal to the joint in all cases with the arms of the goniometer aligned on the finger bones. The DIP, the PIP and MCP joints will be measured in both extension and flexion range of motion. The degrees of measurement will be noted using the neutral-zero method.

SECONDARY OUTCOMES:
Patient satisfaction | Change from baseline to 2, 4 and 8 weeks
  The ICHOM Satisfaction with treatment results questionnaire will be used to assess patient satisfaction. "Treatment" will be replaced by "orthosis" to assess orthotic satisfaction for the 2 and 4 week measurement. To assess satisfaction with treatment outcome, the questionnaire will be used in its original form
Patient Specific Functional Scale (PSFS) | Change from baseline to 4 and 8 weeks
  To measure activity performance and satisfaction with the performance, the investigators will use the Patient Specific Functional Scale (PSFS). The PSFS is a patient specific and activity based short questionnaire where patients must name up to five activities that are currently difficult to do because of the motion limitations in the PIPJ, and give a score from 0-10. At follow-up, patients just must rescore the activities. The total of the scores is then summed up and divided by the numbers of given activities, which is the total score. The difference is considered significant if there is a change of minimum two points for individual activities or of three points for the total score. The PSFS is a reliable, valid, and responsive tool for measuring outcomes in patients with upper extremity issues.
Orthosis diary | continuous
  To monitor adherence with the orthotic intervention, the investigators will give the participants an orthosis diary, where they will note their total orthosis wearing time, whether they were satisfied with their hand performance while wearing the orthosis and when during the day they have been wearing the orthosis. Additionally, the perceived level of pain at rest and while moving before and after the dedicated orthosis wearing time of 6-12 hours per day will be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
We do not plan to publish our results in ICMJE journals.

REFERENCES:
- [Background] Glasgow C, Fleming J, Tooth LR, Peters S. Randomized controlled trial of daily total end range time (TERT) for Capener splinting of the stiff proximal interphalangeal joint. Am J Occup Ther. 2012 Mar-Apr;66(2):243-8. doi: 10.5014/ajot.2012.002816. PMID 22394534
- [Background] Horn KK, Jennings S, Richardson G, Vliet DV, Hefford C, Abbott JH. The patient-specific functional scale: psychometrics, clinimetrics, and application as a clinical outcome measure. J Orthop Sports Phys Ther. 2012 Jan;42(1):30-42. doi: 10.2519/jospt.2012.3727. Epub 2011 Oct 25. PMID 22031594
- [Background] Hefford C, Abbott JH, Arnold R, Baxter GD. The patient-specific functional scale: validity, reliability, and responsiveness in patients with upper extremity musculoskeletal problems. J Orthop Sports Phys Ther. 2012 Feb;42(2):56-65. doi: 10.2519/jospt.2012.3953. Epub 2012 Feb 1. PMID 22333510
- [Background] Schreuders TA. The quadriga phenomenon: a review and clinical relevance. J Hand Surg Eur Vol. 2012 Jul;37(6):513-22. doi: 10.1177/1753193411430810. Epub 2011 Dec 14. PMID 22170246
- [Background] Shaw AV, Verma Y, Tucker S, Jain A, Furniss D. Relative motion orthoses for early active motion after finger extensor and flexor tendon repairs: A systematic review. J Hand Ther. 2023 Apr-Jun;36(2):332-346. doi: 10.1016/j.jht.2023.02.011. Epub 2023 Apr 8. PMID 37037728
- [Background] Arslan OB, Sigirtmac IC, Ayvali C, Bas CE, Ayhan E, Bilgin SS, Oksuz C. The Use of Relative Motion Flexion Orthoses for Chronic Boutonniere Deformity. J Hand Surg Am. 2024 May;49(5):488.e1-488.e8. doi: 10.1016/j.jhsa.2022.08.007. Epub 2022 Oct 4. PMID 36202676
- [Background] Yates SE, Glinsky JV, Hirth MJ, Fuller JT. The use of exercise relative motion orthoses to improve proximal interphalangeal joint motion: A survey of Australian hand therapy practice. J Hand Ther. 2023 Apr-Jun;36(2):414-424. doi: 10.1016/j.jht.2022.12.002. Epub 2023 Apr 6. PMID 37031058
- [Background] Arslan OB, Sahin Y, Sigirtmac IC, Yildiz B, Ayhan E, Oksuz C. Use of relative motion orthoses from the perspective of hand-injured patients: A qualitative study. J Hand Ther. 2023 Apr-Jun;36(2):425-432. doi: 10.1016/j.jht.2023.02.003. Epub 2023 Apr 8. PMID 37037730
- [Background] Howell JW, Ewald SG, Schwartz DA. Exercise relative motion orthoses: Use of the pencil test and variations of its use for assessing and managing different finger conditions. J Hand Ther. 2023 Apr-Jun;36(2):473-478. doi: 10.1016/j.jht.2022.10.004. Epub 2023 Mar 11. No abstract available. PMID 36914489
- [Background] Wajon S, Howell JW. Prescription of exercise relative motion orthoses to improve limited proximal interphalangeal joint movement: A prospective, multi-center, consecutive case series. J Hand Ther. 2023 Apr-Jun;36(2):378-388. doi: 10.1016/j.jht.2021.09.006. Epub 2022 Jan 14. PMID 35039211
- [Background] Michlovitz SL, Harris BA, Watkins MP. Therapy interventions for improving joint range of motion: A systematic review. J Hand Ther. 2004 Apr-Jun;17(2):118-31. doi: 10.1197/j.jht.2004.02.002. PMID 15162100
- [Background] Yates SE, Glinsky JV, Hirth MJ, Fuller JT. Orthotic interventions for restoring proximal interphalangeal joint motion for patients with hand injuries or conditions: A systematic review and meta-analysis. J Hand Ther. 2024 Oct-Dec;37(4):495-506. doi: 10.1016/j.jht.2023.12.018. Epub 2024 Jan 26. PMID 38278697
- [Background] Kamnerdnakta S, Huetteman HE, Chung KC. Complications of Proximal Interphalangeal Joint Injuries: Prevention and Treatment. Hand Clin. 2018 May;34(2):267-288. doi: 10.1016/j.hcl.2017.12.014. PMID 29625645